CLINICAL TRIAL: NCT00482924
Title: Study for the Investigation of New Individual Risk Profiles and Therapeutic Strategies in Obesity Related Cardiovascular and Metabolic Disorders.
Brief Title: Observational Study of Early Metabolic and Vascular Changes in Obesity
Acronym: STYJOBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: Zukunftsfonds Steiermark (Other); Bundesministerium für Gesundheit, Familie und Jugend (Unknown); Steiermärkische Landesregierung (Unknown); Graz University of Technology (Other); University of Graz (Other); Paracelsus Medical University (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harald Mangge, MD, Professor Dr.med., Medical University of Graz
Other Study IDs: A2720000021
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Obesity; Atherosclerosis; Inflammation; Adiponectin Deficiency; Fatty Liver
Keywords: obesity; cardiovascular risk profiles; adipokines; preatherosclerosis; low grade inflammation; dyslipidemia; insulin resistance; brown adipose tissue; white adipose tissue
MeSH Terms: conditions — Obesity; Atherosclerosis; Inflammation; Hypoadiponectinemia; Fatty Liver; Dyslipidemias; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of fasted blood samples between 9 and 12 AM.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Overweight/obese: The cohort consists of age and sex matched normal weighted controls and overweight/obese persons.
  Definition for "overweight": BMI >90th and <97th percentile, if under 18 years of age, and BMI >25 and <29.9 kg/m2 if over 18 years of age.
  Definition for "obese": BMI >97th percentile, if under 18 years of age, and BMI >30kg/m2, if over 18 years of age.
  Interventions: Other: Lifestyle intervention
- Interventional branch: A lifestyle intervention following a holistic schedule was done in a subgroup of obese juveniles.

INTERVENTIONS:
Other: Lifestyle intervention — Regular sports and dietary advices. Controlled by analysis of laboratory parameters, BMI change and performance diagnostics. No drugs included so far.
  Other Names: lifestyle counseling
  Groups: Overweight/obese

SUMMARY:
To work against the increasing burden of obesity, the STYJOBS / EDECTA (STYrian Juvenile OBesity Study / Early DetECtion of Atherosclerosis) project was started at the Medical University of Graz in 2003. STYJOBS / EDECTA is a prospective, observational study to improve the understanding of atherosclerosis, cardiovascular risk, immune mediated low grade Inflammation, metabolic changes, and general disease propensity in obesity. The investigation of the "non-biased" early phase is strongly focused.

Based on this information, new and effective strategies for preclinical diagnostics and early intervention are of main interest. We seek a better understanding of critical lipid profiles, chronic immune-mediated inflammation, disturbed adipokine balance, critical adipose tissue topography, addiction like behaviour, genetics/epigenetics, early vascular pathology, and fatty liver disease. Interventional branches of study tested a holistic strategy comprehending sports, and lifestyle modification for efficiency. The investigative spectrum of STYJOBS / EDECTA comprehends also non-obese body weight extremes i.e. underweight/anorectic people.

DETAILED DESCRIPTION:
Obesity is dramatically increasing in countries with so called western Lifestyle, whereby juveniles are affected in particular. Atherosclerosis, a major consequence of obesity, starts early in life and results in cardiovascular disease and stroke, the main causes of mortality in industrialized countries. STYJOBS / EDECTA is a prospective, observational study to improve the understanding of obesity associated pathologic conditions by investigation of the "non-biased" early phase.

We aim

To identify "individual metabolic high risk patterns" in obesity by linking lab parameters (adipokines, immune-inflammatory mediators, oxidative "stress" biomarkers, lipoproteins, molecular genetics, epigenetics), individual adipose tissue topography, early vascular damage, life style habits, and clinical data.

The STYJOBS/EDECTA-Database comprehends currently data from 1325 subjects.For each proband 282 variables are available (Clinical, anthropometric, carotis IMT, 82; Laboratory/Biomarkers, 100; Glucose metabolism, liver, kidney function, lipids, oxidative/nitrosative stress, adipokines, gut-brain axis, clotting, Genetic/mitochondrial function/miscellaneous,100), and the results of an early interventional trial by a holistic strategy.

To establish a comprehensive biobank. The STYJOBS/EDECTA-biomaterial resource comprises serum/plasma/DNA left over probes from currently 1256 probands.

EDECTA (Early DEteCTion of Atherosclerosis) extends the STYJOBS Database and Bioresource with normal weight and obese probands aged up to 80 years.

To improve the understanding of craving and addiction like behaviour in obesity (e.g.link insulin resistance - control of hedonic inputs).

Thus, the STYJOBS / EDECTA resource comprises in extendo data and biomaterial specimen from subjects afflicted with the preclinical phase of major sequels of obesity such as insulin resistance, cardiovascular disease, and probably also certain sorts of cancer.

To further improve the understanding of dysbalanced energy expenditure in obesity mitochondrial haplotypes are investigated in cooperation with Dr.Weghuber, Dr.Eder and Prof.Sperl from the Salzburg Paracelsus Private Medical School. All genetic and epigenetic measurements are performed by an anonymous approach (data privacy protection) after careful accreditation by the local ethical committee.

The investigative spectrum of STYJOBS / EDECTA is also extended to underweight/anorectic people. This condition is an attractive biologic "counterpart" to the overweight/obese group. Extremely underweight and anorectic patients are afflicted with profound metabolic abnormalities. Thus, it is interesting to investigate anorexia associated risk profiles in comparison to those found in overweight/obese people. Especially the craving like behaviour and the cardiovascular/"ox"Stress risk will be focused in our investigations.

Further, we investigate the role of tryptophan (TRP) metabolism in context with obesity, immune-mediated inflammation, skewing of T helper cells and mechanisms underlying uncontrolled overeating.

ELIGIBILITY:
Inclusion Criteria:

* general healthy condition except overweightness/obesity, age below 55 years

Exclusion Criteria:

* thyroid dysfunction, infections, chronic diseases (e.g. autoimmune, inflammatory), neoplasia

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Probands are residents of Graz and from the federal state of styria.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2003-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Anthropometric changes(BMI, SAT-Topography, waist/hipCF, waist to height ratio) during intervention | 12 months

SECONDARY OUTCOMES:
Obesity related biomarkers (fasting glucose, insulin, HOMA-index, HbA1c, liver transaminases, inflammatory markers, adipokines, clotting parameters, lipids, oxidative stress markers, Biomarkers related to tryptophan metabolism), performance diagnostics. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Harald Mangge, Prof., MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Clinical Institute for Medical and Chemical Laboratory Diagnosis, Graz, Styria, Austria

REFERENCES:
- [Background] Pilz S, Mangge H, Wellnitz B, Seelhorst U, Winkelmann BR, Tiran B, Boehm BO, Marz W. Adiponectin and mortality in patients undergoing coronary angiography. J Clin Endocrinol Metab. 2006 Nov;91(11):4277-86. doi: 10.1210/jc.2006-0836. Epub 2006 Aug 15. PMID 16912132
- [Background] Murr C, Winklhofer-Roob BM, Schroecksnadel K, Maritschnegg M, Mangge H, Bohm BO, Winkelmann BR, Marz W, Fuchs D. Inverse association between serum concentrations of neopterin and antioxidants in patients with and without angiographic coronary artery disease. Atherosclerosis. 2009 Feb;202(2):543-9. doi: 10.1016/j.atherosclerosis.2008.04.047. Epub 2008 May 15. PMID 18556000
- [Background] Pachler C, Ikeoka D, Plank J, Weinhandl H, Suppan M, Mader JK, Bodenlenz M, Regittnig W, Mangge H, Pieber TR, Ellmerer M. Subcutaneous adipose tissue exerts proinflammatory cytokines after minimal trauma in humans. Am J Physiol Endocrinol Metab. 2007 Sep;293(3):E690-6. doi: 10.1152/ajpendo.00034.2007. Epub 2007 Jun 19. PMID 17578890
- [Background] Pilz S, Mangge H, Obermayer-Pietsch B, Marz W. Visfatin/pre-B-cell colony-enhancing factor: a protein with various suggested functions. J Endocrinol Invest. 2007 Feb;30(2):138-44. doi: 10.1007/BF03347412. PMID 17392604
- [Background] Arnold T, Brandlhofer S, Vrtikapa K, Stangl H, Hermann M, Zwiauer K, Mangge H, Karwautz A, Huemer J, Koller D, Schneider WJ, Strobl W. Effect of obesity on plasma clusterin, [corrected] a proposed modulator of leptin action. Pediatr Res. 2011 Mar;69(3):237-42. doi: 10.1203/PDR.0b013e31820930cb. PMID 21135756
- [Background] Fritsch P, Kleber M, Schlagenhauf A, Laschnik B, Fritsch M, Muntean W, Mangge H, Reinehr T. Normalization of haemostatic alterations in overweight children with weight loss due to lifestyle intervention. Atherosclerosis. 2011 May;216(1):170-3. doi: 10.1016/j.atherosclerosis.2011.01.042. Epub 2011 Feb 2. PMID 21334626
- [Background] Hasija R, Pistorio A, Ravelli A, Demirkaya E, Khubchandani R, Guseinova D, Malattia C, Canhao H, Harel L, Foell D, Wouters C, De Cunto C, Huemer C, Kimura Y, Mangge H, Minetti C, Nordal EB, Philippet P, Garozzo R, Martini A, Ruperto N; Pediatric Rheumatology International Trials Organization. Therapeutic approaches in the treatment of juvenile dermatomyositis in patients with recent-onset disease and in those experiencing disease flare: an international multicenter PRINTO study. Arthritis Rheum. 2011 Oct;63(10):3142-52. doi: 10.1002/art.30475. PMID 21647864
- [Background] Almer G, Wernig K, Saba-Lepek M, Haj-Yahya S, Rattenberger J, Wagner J, Gradauer K, Frascione D, Pabst G, Leitinger G, Mangge H, Zimmer A, Prassl R. Adiponectin-coated nanoparticles for enhanced imaging of atherosclerotic plaques. Int J Nanomedicine. 2011;6:1279-90. doi: 10.2147/IJN.S18739. Epub 2011 Jun 21. PMID 21753879
- [Background] Almer G, Saba-Lepek M, Haj-Yahya S, Rohde E, Strunk D, Frohlich E, Prassl R, Mangge H. Globular domain of adiponectin: promising target molecule for detection of atherosclerotic lesions. Biologics. 2011;5:95-105. doi: 10.2147/BTT.S22863. Epub 2011 Sep 7. PMID 22022204
- [Background] Landauer F, Huber G, Paulmichl K, O'Malley G, Mangge H, Weghuber D. Timely diagnosis of malalignment of the distal extremities is crucial in morbidly obese juveniles. Obes Facts. 2013;6(6):542-51. doi: 10.1159/000357280. Epub 2013 Dec 6. PMID 24335156
- [Background] Reininghaus EZ, McIntyre RS, Reininghaus B, Geisler S, Bengesser SA, Lackner N, Hecht K, Birner A, Kattnig F, Unterweger R, Kapfhammer HP, Zelzer S, Fuchs D, Mangge H. Tryptophan breakdown is increased in euthymic overweight individuals with bipolar disorder: a preliminary report. Bipolar Disord. 2014 Jun;16(4):432-40. doi: 10.1111/bdi.12166. Epub 2013 Dec 12. PMID 24330408
- [Background] Gradauer K, Barthelmes J, Vonach C, Almer G, Mangge H, Teubl B, Roblegg E, Dunnhaupt S, Frohlich E, Bernkop-Schnurch A, Prassl R. Liposomes coated with thiolated chitosan enhance oral peptide delivery to rats. J Control Release. 2013 Dec 28;172(3):872-8. doi: 10.1016/j.jconrel.2013.10.011. Epub 2013 Oct 16. PMID 24140721
- [Background] Bengesser SA, Lackner N, Birner A, Fellendorf FT, Platzer M, Mitteregger A, Unterweger R, Reininghaus B, Mangge H, Wallner-Liebmann SJ, Zelzer S, Fuchs D, McIntyre RS, Kapfhammer HP, Reininghaus EZ. Peripheral markers of oxidative stress and antioxidative defense in euthymia of bipolar disorder--Gender and obesity effects. J Affect Disord. 2015 Feb 1;172:367-74. doi: 10.1016/j.jad.2014.10.014. Epub 2014 Oct 22. PMID 25451439
- [Background] Lackner N, Mangge H, Reininghaus EZ, McIntyre RS, Bengesser SA, Birner A, Reininghaus B, Kapfhammer HP, Wallner-Liebmann SJ. Body fat distribution and associations with metabolic and clinical characteristics in bipolar individuals. Eur Arch Psychiatry Clin Neurosci. 2015 Jun;265(4):313-9. doi: 10.1007/s00406-014-0559-8. Epub 2014 Nov 8. PMID 25381166
- [Background] Mangge H, Becker K, Fuchs D, Gostner JM. Antioxidants, inflammation and cardiovascular disease. World J Cardiol. 2014 Jun 26;6(6):462-77. doi: 10.4330/wjc.v6.i6.462. PMID 24976919
- [Background] Wallner-Liebmann SJ, Moeller R, Horejsi R, Jurimae T, Jurimae J, Maestu J, Purge P, Saar M, Tafeit E, Kaimbacher P, Kruschitz R, Weghuber D, Schnedl WJ, Mangge H. Normal weight estonian prepubertal boys show a more cardiovascular-risk-associated adipose tissue distribution than austrian counterparts. ISRN Obes. 2013 Jan 14;2013:506751. doi: 10.1155/2013/506751. eCollection 2013. PMID 24555148
- [Background] Mangge H, Weghuber D, Prassl R, Haara A, Schnedl W, Postolache TT, Fuchs D. The Role of Vitamin D in Atherosclerosis Inflammation Revisited: More a Bystander than a Player? Curr Vasc Pharmacol. 2015;13(3):392-8. doi: 10.2174/1570161111666131209125454. PMID 24329737
- [Background] Raheja UK, Fuchs D, Giegling I, Brenner LA, Rovner SF, Mohyuddin I, Weghuber D, Mangge H, Rujescu D, Postolache TT. In psychiatrically healthy individuals, overweight women but not men have lower tryptophan levels. Pteridines. 2015 Jun;26(2):79-84. doi: 10.1515/pterid-2015-0002. PMID 26251562
- [Background] Mangge H, Pruller F, Zelzer S, Ainodhofer H, Pailer S, Kieslinger P, Haybaeck J, Obermayer-Pietsch B, Cvirn G, Gruber HJ. Hypothyroidism Exacerbates Thrombophilia in Female Rats Fed with a High Fat Diet. Int J Mol Sci. 2015 Jul 10;16(7):15776-84. doi: 10.3390/ijms160715776. PMID 26184174
- [Background] Lackner N, Bengesser SA, Birner A, Painold A, Fellendorf FT, Platzer M, Reininghaus B, Weiss EM, Mangge H, McIntyre RS, Fuchs D, Kapfhammer HP, Wallner-Liebmann SJ, Reininghaus EZ. Abdominal obesity is associated with impaired cognitive function in euthymic bipolar individuals. World J Biol Psychiatry. 2016 Oct;17(7):535-46. doi: 10.3109/15622975.2015.1046917. Epub 2015 Jun 12. PMID 26068130
- [Background] Zelzer S, Mangge H, Pailer S, Ainoedhofer H, Kieslinger P, Stojakovic T, Scharnagl H, Pruller F, Weghuber D, Datz C, Haybaeck J, Obermayer-Pietsch B, Trummer C, Gostner J, Gruber HJ. Oxidized LDL Is Strictly Limited to Hyperthyroidism Irrespective of Fat Feeding in Female Sprague Dawley Rats. Int J Mol Sci. 2015 May 21;16(5):11689-98. doi: 10.3390/ijms160511689. PMID 26006242
- [Background] Mangge H, Almer G, Stelzer I, Reininghaus E, Prassl R. Laboratory medicine for molecular imaging of atherosclerosis. Clin Chim Acta. 2014 Nov 1;437:19-24. doi: 10.1016/j.cca.2014.06.029. Epub 2014 Jul 5. PMID 25003647
- [Background] Mangge H, Ciardi C, Becker K, Strasser B, Fuchs D, Gostner JM. Influence of Antioxidants on Leptin Metabolism and its Role in the Pathogenesis of Obesity. Adv Exp Med Biol. 2017;960:399-413. doi: 10.1007/978-3-319-48382-5_17. PMID 28585209
- [Background] Mangge H. Beyond Cholesterol - New Cardiovascular Biomarkers. Nestle Nutr Inst Workshop Ser. 2016;84:81-8. doi: 10.1159/000436990. Epub 2016 Jan 14. PMID 26764476
- [Result] Moeller R, Horejsi R, Pilz S, Lang N, Sargsyan K, Dimitrova R, Tafeit E, Giuliani A, Almer G, Mangge H. Evaluation of risk profiles by subcutaneous adipose tissue topography in obese juveniles. Obesity (Silver Spring). 2007 May;15(5):1319-24. doi: 10.1038/oby.2007.154. PMID 17495209
- [Result] Cimenti C, Mangge H, Haidl H, Zach D, Muntean W. Thrombin generation in severely obese children. J Thromb Haemost. 2006 Aug;4(8):1834-6. doi: 10.1111/j.1538-7836.2006.02038.x. No abstract available. PMID 16879229
- [Result] Pilz S, Horejsi R, Moller R, Almer G, Scharnagl H, Stojakovic T, Dimitrova R, Weihrauch G, Borkenstein M, Maerz W, Schauenstein K, Mangge H. Early atherosclerosis in obese juveniles is associated with low serum levels of adiponectin. J Clin Endocrinol Metab. 2005 Aug;90(8):4792-6. doi: 10.1210/jc.2005-0167. Epub 2005 May 31. PMID 15928248
- [Result] Mangge H, Schauenstein K, Stroedter L, Griesl A, Maerz W, Borkenstein M. Low grade inflammation in juvenile obesity and type 1 diabetes associated with early signs of atherosclerosis. Exp Clin Endocrinol Diabetes. 2004 Jul;112(7):378-82. doi: 10.1055/s-2004-821023. PMID 15239023
- [Result] Gruber HJ, Mayer C, Meinitzer A, Almer G, Horejsi R, Moller R, Pilz S, Marz W, Gasser R, Truschnig-Wilders M, Mangge H. Asymmetric dimethylarginine (ADMA) is tightly correlated with growth in juveniles without correlations to obesity related disorders. Exp Clin Endocrinol Diabetes. 2008 Oct;116(9):520-4. doi: 10.1055/s-2008-1062712. Epub 2008 Apr 1. PMID 18523919
- [Result] Mangge H, Pilz S, Haj-Yahya S, Almer G. Uric acid indicates a high cardiovascular risk profile but is not closely associated with insulin resistance in obese adolescents. Diabetes Care. 2008 Apr;31(4):e21. doi: 10.2337/dc07-2411. No abstract available. PMID 18375422
- [Result] Gruber HJ, Mayer C, Mangge H, Fauler G, Grandits N, Wilders-Truschnig M. Obesity reduces the bioavailability of nitric oxide in juveniles. Int J Obes (Lond). 2008 May;32(5):826-31. doi: 10.1038/sj.ijo.0803795. Epub 2008 Jan 15. PMID 18197180
- [Result] Mangge H, Almer G, Haj-Yahya S, Grandits N, Gasser R, Pilz S, Moller R, Horejsi R. Nuchal thickness of subcutaneous adipose tissue is tightly associated with an increased LMW/total adiponectin ratio in obese juveniles. Atherosclerosis. 2009 Mar;203(1):277-83. doi: 10.1016/j.atherosclerosis.2008.06.013. Epub 2008 Jun 26. PMID 18656877
- [Result] Wilders-Truschnig M, Mangge H, Lieners C, Gruber H, Mayer C, Marz W. IgG antibodies against food antigens are correlated with inflammation and intima media thickness in obese juveniles. Exp Clin Endocrinol Diabetes. 2008 Apr;116(4):241-5. doi: 10.1055/s-2007-993165. Epub 2007 Dec 10. PMID 18072008
- [Result] Mangge H, Almer G, Haj-Yahya S, Pilz S, Gasser R, Moller R, Horejsi R. Preatherosclerosis and adiponectin subfractions in obese adolescents. Obesity (Silver Spring). 2008 Dec;16(12):2578-84. doi: 10.1038/oby.2008.439. Epub 2008 Oct 9. PMID 18846045
- [Result] Wallner-Liebmann S, Koschutnig K, Reishofer G, Sorantin E, Blaschitz B, Kruschitz R, Unterrainer HF, Gasser R, Freytag F, Bauer-Denk C, Schienle A, Schafer A, Mangge H. Insulin and hippocampus activation in response to images of high-calorie food in normal weight and obese adolescents. Obesity (Silver Spring). 2010 Aug;18(8):1552-7. doi: 10.1038/oby.2010.26. Epub 2010 Feb 18. PMID 20168310
- [Result] Mangge H, Freytag F, Almer G, Weghuber D, Bauer-Denk C, Fuchs D. Serum neopterin is not increased in obese juveniles. J Obes. 2011;2011:946795. doi: 10.1155/2011/946795. Epub 2011 Jan 12. PMID 21274279
- [Result] Mangge H, Almer G, Truschnig-Wilders M, Schmidt A, Gasser R, Fuchs D. Inflammation, adiponectin, obesity and cardiovascular risk. Curr Med Chem. 2010;17(36):4511-20. doi: 10.2174/092986710794183006. PMID 21062254
- [Result] Mangge H, Renner W, Almer G, Weghuber D, Moller R, Horejsi R. Rs9939609 variant of the fat mass and obesity-associated gene and trunk obesity in adolescents. J Obes. 2011;2011:186368. doi: 10.1155/2011/186368. Epub 2011 Jan 13. PMID 21318054
- [Result] Mangge H, Almer G, Zelzer S, Vasan R, Kraigher-Krainer E, Gasser R, Schnedl W, Ille R, Wallner S, Moller R, Horejsi R, Weghuber D. N-terminal pro-B-type natriuretic peptide in early and advanced phases of obesity. Clin Chem Lab Med. 2011 Sep;49(9):1539-45. doi: 10.1515/CCLM.2011.627. Epub 2011 Jun 10. PMID 21663466
- [Result] Zelzer S, Fuchs N, Almer G, Raggam RB, Pruller F, Truschnig-Wilders M, Schnedl W, Horejsi R, Moller R, Weghuber D, Ille R, Mangge H. High density lipoprotein cholesterol level is a robust predictor of lipid peroxidation irrespective of gender, age, obesity, and inflammatory or metabolic biomarkers. Clin Chim Acta. 2011 Jul 15;412(15-16):1345-9. doi: 10.1016/j.cca.2011.03.031. Epub 2011 Apr 15. PMID 21515245
- [Result] Stelzer I, Zelzer S, Raggam RB, Pruller F, Truschnig-Wilders M, Meinitzer A, Schnedl WJ, Horejsi R, Moller R, Weghuber D, Reeves G, Postolache TT, Mangge H. Link between leptin and interleukin-6 levels in the initial phase of obesity related inflammation. Transl Res. 2012 Feb;159(2):118-24. doi: 10.1016/j.trsl.2011.10.001. Epub 2011 Nov 4. PMID 22243796
- [Result] Pruller F, Raggam RB, Posch V, Almer G, Truschnig-Wilders M, Horejsi R, Moller R, Weghuber D, Ille R, Schnedl W, Mangge H. Trunk weighted obesity, cholesterol levels and low grade inflammation are main determinants for enhanced thrombin generation. Atherosclerosis. 2012 Jan;220(1):215-8. doi: 10.1016/j.atherosclerosis.2011.09.035. Epub 2011 Oct 14. PMID 22035573
- [Result] Mangge H, Summers KL, Meinitzer A, Zelzer S, Almer G, Prassl R, Schnedl WJ, Reininghaus E, Paulmichl K, Weghuber D, Fuchs D. Obesity-related dysregulation of the tryptophan-kynurenine metabolism: role of age and parameters of the metabolic syndrome. Obesity (Silver Spring). 2014 Jan;22(1):195-201. doi: 10.1002/oby.20491. Epub 2013 Jul 5. PMID 23625535
- [Result] Mangge H, Summers K, Almer G, Prassl R, Weghuber D, Schnedl W, Fuchs D. Antioxidant food supplements and obesity-related inflammation. Curr Med Chem. 2013;20(18):2330-7. doi: 10.2174/0929867311320180004. PMID 23531214
- [Result] Weghuber D, Zelzer S, Stelzer I, Paulmichl K, Kammerhofer D, Schnedl W, Molnar D, Mangge H. High risk vs. "metabolically healthy" phenotype in juvenile obesity - neck subcutaneous adipose tissue and serum uric acid are clinically relevant. Exp Clin Endocrinol Diabetes. 2013 Jul;121(7):384-90. doi: 10.1055/s-0033-1341440. Epub 2013 Mar 21. PMID 23519645
- [Result] Mangge H, Zelzer S, Puerstner P, Schnedl WJ, Reeves G, Postolache TT, Weghuber D. Uric acid best predicts metabolically unhealthy obesity with increased cardiovascular risk in youth and adults. Obesity (Silver Spring). 2013 Jan;21(1):E71-7. doi: 10.1002/oby.20061. Epub 2013 Jan 29. PMID 23401248
- [Result] Almer G, Frascione D, Pali-Scholl I, Vonach C, Lukschal A, Stremnitzer C, Diesner SC, Jensen-Jarolim E, Prassl R, Mangge H. Interleukin-10: an anti-inflammatory marker to target atherosclerotic lesions via PEGylated liposomes. Mol Pharm. 2013 Jan 7;10(1):175-86. doi: 10.1021/mp300316n. Epub 2012 Dec 4. PMID 23176185
- [Result] Mangge H, Zelzer S, Meinitzer A, Stelzer I, Schnedl WJ, Weghuber D, Fuchs D, Postolache TT, Aigner E, Datz C, Reininghaus EZ. 25OH-Vitamin D3 Levels in Obesity and Metabolic Syndrome-Unaltered in Young and not Correlated to Carotid IMT in All Ages. Curr Pharm Des. 2015;21(17):2243-9. doi: 10.2174/1381612821666150105160931. PMID 25557634
- [Result] Mangge H, Stelzer I, Reininghaus EZ, Weghuber D, Postolache TT, Fuchs D. Disturbed tryptophan metabolism in cardiovascular disease. Curr Med Chem. 2014 Jun;21(17):1931-7. doi: 10.2174/0929867321666140304105526. PMID 24606499
- [Result] Ebner S, Mangge H, Langhof H, Halle M, Siegrist M, Aigner E, Paulmichl K, Paulweber B, Datz C, Sperl W, Kofler B, Weghuber D. Mitochondrial Haplogroup T Is Associated with Obesity in Austrian Juveniles and Adults. PLoS One. 2015 Aug 31;10(8):e0135622. doi: 10.1371/journal.pone.0135622. eCollection 2015. PMID 26322975
- [Result] Mangge H, Baumgartner B, Schnedl W. Letter: PNPLA3, metabolic syndrome and NAFLD status in obese subjects--authors' reply. Aliment Pharmacol Ther. 2015 Sep;42(5):630-1. doi: 10.1111/apt.13318. No abstract available. PMID 26238581
- [Result] Mangge H, Baumgartner BG, Zelzer S, Pruller F, Schnedl WJ, Reininghaus EZ, Haybaeck J, Lackner C, Stauber R, Aigner E, Weghuber D. Patatin-like phospholipase 3 (rs738409) gene polymorphism is associated with increased liver enzymes in obese adolescents and metabolic syndrome in all ages. Aliment Pharmacol Ther. 2015 Jul;42(1):99-105. doi: 10.1111/apt.13232. Epub 2015 May 5. PMID 25939720
- [Result] Mangge H, Zelzer S, Pruller F, Schnedl WJ, Weghuber D, Enko D, Bergsten P, Haybaeck J, Meinitzer A. Branched-chain amino acids are associated with cardiometabolic risk profiles found already in lean, overweight and obese young. J Nutr Biochem. 2016 Jun;32:123-7. doi: 10.1016/j.jnutbio.2016.02.007. Epub 2016 Mar 21. PMID 27142745
- [Result] Marsche G, Zelzer S, Meinitzer A, Kern S, Meissl S, Pregartner G, Weghuber D, Almer G, Mangge H. Adiponectin Predicts High-Density Lipoprotein Cholesterol Efflux Capacity in Adults Irrespective of Body Mass Index and Fat Distribution. J Clin Endocrinol Metab. 2017 Nov 1;102(11):4117-4123. doi: 10.1210/jc.2017-00933. PMID 28938424
- [Derived] Mangge H, Renner W, Almer G, Gruber HJ, Zelzer S, Moeller R, Horejsi R, Herrmann M. Subcutaneous adipose tissue distribution and telomere length. Clin Chem Lab Med. 2019 Aug 27;57(9):1358-1363. doi: 10.1515/cclm-2018-0801. PMID 30913032